CLINICAL TRIAL: NCT05216614
Title: Fluvoxamine to Augment Olfactory Recovery For Long COVID-19 Parosmia (FluCOP Trial)
Brief Title: Fluvoxamine to Augment Olfactory Recovery For Long COVID-19 Parosmia
Acronym: FluCOP
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Unable to obtain investigational product
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 202111124
Record Dates: First submitted 2022-01-24; First posted 2022-01-31 (Actual); Last update posted 2022-03-11 (Actual); Status verified 2022-02

CONDITIONS: COVID-19; Olfactory Disorder; Parosmia
MeSH Terms: conditions — COVID-19; Olfaction Disorders | interventions — Fluvoxamine

STUDY DESIGN:
Intervention Model Description: Double-blinded, randomized, placebo-controlled trial
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: double-blinded, both participants and investigators will be blinded. Intervention will be packaged in blinded fashion by pharmacist before being shipped to participants by research assistant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Fluvoxamine (Experimental): This arm will be given the active treatment, oral fluvoxamine capsules of 25 mg each.
  The first six weeks will be gradual titration (weeks 1 & 2 25mg BID, weeks 3 & 4 75mg BID, weeks 5 & 6 100mg BID).
  The following six weeks will be fixed dose of 100mg TID.
  The last two weeks will be a taper down (first week 50mg BID and second week 25mg BID)
  There will be 14 weeks of active treatment and assessments will be conducted after completion of week 12, prior to beginning taper down period.
  Interventions: Drug: Fluvoxamine
- Placebo (Placebo Comparator): Placebo capsules that look, smell, and taste like fluvoxamine capsules will be given to the placebo arm.
  To preserve double-blinding of the study, subjects will receive one capsule BID during the first six weeks following the titration schedule and one capsule TID during the next six weeks for the fixed-dose period.
  Subjects will then taper-down placebo to imitate the fluvoxamine arm for two weeks.
  Assessments will be conducted at 12 weeks following completion of fixed-dose period, prior to starting taper down period.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Fluvoxamine — Fluvoxamine is an SSRI used for depression and anxiety disorders. This study will investigate the efficacy of fluvoxamine for improvement of olfactory dysfunction in subjects with post-Covid-19 parosmia.
  Other Names: Luvox
  Arms: Fluvoxamine
Drug: Placebo — lactose placebo capsules identical to fluvoxamine capsules in order to preserve blind
  Arms: Placebo

SUMMARY:
This study will investigate the efficacy of oral fluvoxamine in olfactory improvement following Covid-19- associated parosmia. This is a randomized, double-blinded, placebo-controlled trial.

DETAILED DESCRIPTION:
The drug will be given over a 14 weeks with six weeks titrating up, six weeks maintaining highest dose, and up to two weeks tapering down. Assessments will be collected following week 12 to measure change in olfactory function from baseline between the two study groups.

ELIGIBILITY:
Inclusion Criteria:

* Men and women between the ages 18 to 70 years
* Residing within the states of Missouri or Illinois
* Complaints of odors of certain things or everything are distorted
* Olfactory dysfunction that has persisted for >2 months after suspected COVID-19 infection
* Ability to read, write, and understand English

Exclusion Criteria:

* History of olfactory dysfunction prior to COVID-19 infection
* Any use of concomitant therapies specifically for the treatment of olfactory dysfunction
* History of olfactory dysfunction of longer than 12 months
* History of bipolar disorder as SSRIs can theoretically destabilize bipolar disorder
* Participants with symptoms of depression as evidenced by a score of 10 or greater on the Patient Health Questionnaire-9 (PHQ-9).95 The PHQ-9 is a nine-item questionnaire designed to assess and aid in diagnosing patients with depression in clinical and community settings.
* History of neurodegenerative disease (i.e., Alzheimer's dementia, Parkinson's disease, Lewy body dementia, frontotemporal dementia)
* History of chronic rhinosinusitis or sinus surgery
* Pregnant or breastfeeding mothers.
* Already enrolled in another COVID 19 medication trial or receipt of monoclonal antibody infusion.
* Taking donepezil or fluoxetine (rationale: these drugs are S1R agonists) or sertraline (a S1R antagonist).
* Participants taking theophylline, tizanidine, clozapine, or olanzapine (drugs with a narrow therapeutic index that are primarily metabolized by CYP 1A2, which is inhibited by fluvoxamine.
* Taking another SSRI, unless at a low dose (e.g., escitalopram 5mg) such that adding fluvoxamine would not put patient at risk for serotonin syndrome.
* Taking coumadin based on theoretical risk of increased bleeding with fluvoxamine.
* Unable to provide informed consent.
* Unable to perform the study procedures.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-12-14 (Actual); Primary Completion 2022-02-22 (Actual); Study Completion 2022-02-22 (Actual)

PRIMARY OUTCOMES:
Clinical Global Impression Scale (CGI) | CGI-S and CGI-P will be administered at Baseline and Week 12 after completion of fixed-dose period, prior to taper down, to measure change. CGI-I will be administered at Week 12 after completion of fixed-dose period, prior to taper down
  The CGI has two components - the CGI-Severity and the CGI-Improvement.
  Scores on the CGI-Severity Scale range from 1 to 7 (1 is Normal, 7 is Complete loss of smell) and provide information on the patient's perceived severity of their dysfunction at baseline. The score on the CGI-Improvement Scale ranges from 1 to 7 (1 is Very Much Improved, 7 is Very Much Worsened). Each rating is well defined to maximize accuracy. Participants reporting 3 as Minimally Improved, 2 as Much Improved, or 1 as Very Much Improved in the CGI-I will be deemed responders to treatment, and the number of responders to non-responders will be compared between the two arms.
  The Clinical Global Impression-Severity Scale for Parosmia (CGI-P) will also be used. The CGI-P Scale ranges from 1 to 5, where 1 is No Distortion, 2 is Mild Distortion, 3 is Moderate Distortion, 4 is Mostly Distorted, and 5 is Complete Distortion.

SECONDARY OUTCOMES:
University of Pennsylvania Smell Identification Test (UPSIT) | Baseline and Week 12 after completion of fixed-dose period, prior to taper down, to measure change from baseline
  The UPSIT is composed of 40 strips of microencapsulated odorants, which are present on the bottom of each page, just below a four-alternative multiple-choice question. For a given item, the patient releases an odor by scratching the microencapsulated pad with a pencil tip, smells the pad, and indicates the odor quality from four alternatives. Even if no smell is perceived, a response is required (i.e., the test is forced-choice). The subject's total correct score out of the 40 items is determined and provides an objective measure of olfactory function.
Olfactory Dysfunction Outcomes Rating (ODOR) | Baseline and Week 12 after completion of fixed-dose period, prior to taper down, to measure change from baseline
  The ODOR questionnaire is a 28-item disease-specific health status survey to assess the physical problems, functional impairments, and emotional consequences secondary to olfactory dysfunction. ODOR was developed and validated by Dr. Jake Lee and colleagues in the Clinical Outcomes Research Office at Washington University
The Depression, Anxiety and Stress Scale - 21 Items (DASS-21) | Baseline and Week 12 after completion of fixed-dose period, prior to taper down, to measure change from baseline
  The DASS-21 is a set of three self-report scales designed to measure the emotional state of depression, anxiety, and stress. Each of the three DASS-21 scales contains 7 items, divided into subscales with similar content. The depression scale assesses dysphoria, hopelessness, devaluation of life, self-deprecation, lack of interest / involvement, anhedonia and inertia. The anxiety scale assesses autonomic arousal, skeletal muscle effects, situational anxiety, and subjective experience of anxious affect. The stress scale is sensitive to levels of chronic non- specific arousal and assesses difficulty relaxing, nervous arousal, and being easily upset / agitated, irritable / over-reactive and impatient. Scores for depression, anxiety and stress are calculated by summing the scores for the relevant items.
The Smell Catastrophizing Scale (SCS) | Baseline and Week 12 after completion of fixed-dose period, prior to taper down, to measure change from baseline
  The SCS is a 13-item scale that asks the participants to describe the degree to which they have specific thoughts and feelings as a result of their sense of smell problems.
36-Item Short Form Health Survey (SF-36) | Baseline and Week 12 after completion of fixed-dose period, prior to taper down, to measure change from baseline
  The SF-36 is a 36-item questionnaire evaluating physical functioning, bodily pain, role limitations due to physical health problems, role limitations due to personal or emotional problems, emotional well-being, social functioning, energy/fatigue, and general health perceptions. This test allows us to study the general health overall quality of life changes for those suffering from COVID-19 related OD.

CONTACTS AND LOCATIONS:
Overall Officials: Jay F Piccirillo, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lechien JR, Chiesa-Estomba CM, De Siati DR, Horoi M, Le Bon SD, Rodriguez A, Dequanter D, Blecic S, El Afia F, Distinguin L, Chekkoury-Idrissi Y, Hans S, Delgado IL, Calvo-Henriquez C, Lavigne P, Falanga C, Barillari MR, Cammaroto G, Khalife M, Leich P, Souchay C, Rossi C, Journe F, Hsieh J, Edjlali M, Carlier R, Ris L, Lovato A, De Filippis C, Coppee F, Fakhry N, Ayad T, Saussez S. Olfactory and gustatory dysfunctions as a clinical presentation of mild-to-moderate forms of the coronavirus disease (COVID-19): a multicenter European study. Eur Arch Otorhinolaryngol. 2020 Aug;277(8):2251-2261. doi: 10.1007/s00405-020-05965-1. Epub 2020 Apr 6. PMID 32253535
- [Background] Wang D, Hu B, Hu C, Zhu F, Liu X, Zhang J, Wang B, Xiang H, Cheng Z, Xiong Y, Zhao Y, Li Y, Wang X, Peng Z. Clinical Characteristics of 138 Hospitalized Patients With 2019 Novel Coronavirus-Infected Pneumonia in Wuhan, China. JAMA. 2020 Mar 17;323(11):1061-1069. doi: 10.1001/jama.2020.1585. PMID 32031570
- [Background] Huang C, Wang Y, Li X, Ren L, Zhao J, Hu Y, Zhang L, Fan G, Xu J, Gu X, Cheng Z, Yu T, Xia J, Wei Y, Wu W, Xie X, Yin W, Li H, Liu M, Xiao Y, Gao H, Guo L, Xie J, Wang G, Jiang R, Gao Z, Jin Q, Wang J, Cao B. Clinical features of patients infected with 2019 novel coronavirus in Wuhan, China. Lancet. 2020 Feb 15;395(10223):497-506. doi: 10.1016/S0140-6736(20)30183-5. Epub 2020 Jan 24. PMID 31986264
- [Background] Zhu N, Zhang D, Wang W, Li X, Yang B, Song J, Zhao X, Huang B, Shi W, Lu R, Niu P, Zhan F, Ma X, Wang D, Xu W, Wu G, Gao GF, Tan W; China Novel Coronavirus Investigating and Research Team. A Novel Coronavirus from Patients with Pneumonia in China, 2019. N Engl J Med. 2020 Feb 20;382(8):727-733. doi: 10.1056/NEJMoa2001017. Epub 2020 Jan 24. PMID 31978945
- [Background] Guan WJ, Ni ZY, Hu Y, Liang WH, Ou CQ, He JX, Liu L, Shan H, Lei CL, Hui DSC, Du B, Li LJ, Zeng G, Yuen KY, Chen RC, Tang CL, Wang T, Chen PY, Xiang J, Li SY, Wang JL, Liang ZJ, Peng YX, Wei L, Liu Y, Hu YH, Peng P, Wang JM, Liu JY, Chen Z, Li G, Zheng ZJ, Qiu SQ, Luo J, Ye CJ, Zhu SY, Zhong NS; China Medical Treatment Expert Group for Covid-19. Clinical Characteristics of Coronavirus Disease 2019 in China. N Engl J Med. 2020 Apr 30;382(18):1708-1720. doi: 10.1056/NEJMoa2002032. Epub 2020 Feb 28. PMID 32109013
- [Background] Yang X, Yu Y, Xu J, Shu H, Xia J, Liu H, Wu Y, Zhang L, Yu Z, Fang M, Yu T, Wang Y, Pan S, Zou X, Yuan S, Shang Y. Clinical course and outcomes of critically ill patients with SARS-CoV-2 pneumonia in Wuhan, China: a single-centered, retrospective, observational study. Lancet Respir Med. 2020 May;8(5):475-481. doi: 10.1016/S2213-2600(20)30079-5. Epub 2020 Feb 24. PMID 32105632
- [Background] Zhou F, Yu T, Du R, Fan G, Liu Y, Liu Z, Xiang J, Wang Y, Song B, Gu X, Guan L, Wei Y, Li H, Wu X, Xu J, Tu S, Zhang Y, Chen H, Cao B. Clinical course and risk factors for mortality of adult inpatients with COVID-19 in Wuhan, China: a retrospective cohort study. Lancet. 2020 Mar 28;395(10229):1054-1062. doi: 10.1016/S0140-6736(20)30566-3. Epub 2020 Mar 11. PMID 32171076
- [Background] Jafek BW, Murrow B, Michaels R, Restrepo D, Linschoten M. Biopsies of human olfactory epithelium. Chem Senses. 2002 Sep;27(7):623-8. doi: 10.1093/chemse/27.7.623. PMID 12200342
- [Background] Gudziol V, Buschhuter D, Abolmaali N, Gerber J, Rombaux P, Hummel T. Increasing olfactory bulb volume due to treatment of chronic rhinosinusitis--a longitudinal study. Brain. 2009 Nov;132(Pt 11):3096-101. doi: 10.1093/brain/awp243. Epub 2009 Sep 22. PMID 19773353
- [Background] Schwob JE. Neural regeneration and the peripheral olfactory system. Anat Rec. 2002 Feb 15;269(1):33-49. doi: 10.1002/ar.10047. PMID 11891623
- [Background] Brann JH, Firestein SJ. A lifetime of neurogenesis in the olfactory system. Front Neurosci. 2014 Jun 26;8:182. doi: 10.3389/fnins.2014.00182. eCollection 2014. PMID 25018692
- [Background] Hoffman HJ, Rawal S, Li CM, Duffy VB. New chemosensory component in the U.S. National Health and Nutrition Examination Survey (NHANES): first-year results for measured olfactory dysfunction. Rev Endocr Metab Disord. 2016 Jun;17(2):221-40. doi: 10.1007/s11154-016-9364-1. PMID 27287364
- [Background] Liu B, Luo Z, Pinto JM, Shiroma EJ, Tranah GJ, Wirdefeldt K, Fang F, Harris TB, Chen H. Relationship Between Poor Olfaction and Mortality Among Community-Dwelling Older Adults: A Cohort Study. Ann Intern Med. 2019 May 21;170(10):673-681. doi: 10.7326/M18-0775. Epub 2019 Apr 30. PMID 31035288
- [Background] Pinto JM, Wroblewski KE, Kern DW, Schumm LP, McClintock MK. Olfactory dysfunction predicts 5-year mortality in older adults. PLoS One. 2014 Oct 1;9(10):e107541. doi: 10.1371/journal.pone.0107541. eCollection 2014. PMID 25271633
- [Background] Van Regemorter V, Hummel T, Rosenzweig F, Mouraux A, Rombaux P, Huart C. Mechanisms Linking Olfactory Impairment and Risk of Mortality. Front Neurosci. 2020 Feb 21;14:140. doi: 10.3389/fnins.2020.00140. eCollection 2020. PMID 32153360
- [Background] Soler ZM, Patel ZM, Turner JH, Holbrook EH. A primer on viral-associated olfactory loss in the era of COVID-19. Int Forum Allergy Rhinol. 2020 Jul;10(7):814-820. doi: 10.1002/alr.22578. Epub 2020 Jun 1. PMID 32271490
- [Background] Bitter T, Gudziol H, Burmeister HP, Mentzel HJ, Guntinas-Lichius O, Gaser C. Anosmia leads to a loss of gray matter in cortical brain areas. Chem Senses. 2010 Jun;35(5):407-15. doi: 10.1093/chemse/bjq028. Epub 2010 Mar 15. PMID 20231262
- [Background] Pekala K, Chandra RK, Turner JH. Efficacy of olfactory training in patients with olfactory loss: a systematic review and meta-analysis. Int Forum Allergy Rhinol. 2016 Mar;6(3):299-307. doi: 10.1002/alr.21669. Epub 2015 Dec 1. PMID 26624966
- [Background] Murphy MP, Fishman P, Short SO, Sullivan SD, Yueh B, Weymuller EA Jr. Health care utilization and cost among adults with chronic rhinosinusitis enrolled in a health maintenance organization. Otolaryngol Head Neck Surg. 2002 Nov;127(5):367-76. doi: 10.1067/mhn.2002.129815. PMID 12447229
- [Background] Schiffman SS, Warwick ZS. Flavor enhancement of foods for the elderly can reverse anorexia. Neurobiol Aging. 1988 Jan-Feb;9(1):24-6. doi: 10.1016/s0197-4580(88)80009-5. PMID 3164095
- [Background] Sungnak W, Huang N, Becavin C, Berg M, Queen R, Litvinukova M, Talavera-Lopez C, Maatz H, Reichart D, Sampaziotis F, Worlock KB, Yoshida M, Barnes JL; HCA Lung Biological Network. SARS-CoV-2 entry factors are highly expressed in nasal epithelial cells together with innate immune genes. Nat Med. 2020 May;26(5):681-687. doi: 10.1038/s41591-020-0868-6. Epub 2020 Apr 23. PMID 32327758
- [Background] Rockx B, Kuiken T, Herfst S, Bestebroer T, Lamers MM, Oude Munnink BB, de Meulder D, van Amerongen G, van den Brand J, Okba NMA, Schipper D, van Run P, Leijten L, Sikkema R, Verschoor E, Verstrepen B, Bogers W, Langermans J, Drosten C, Fentener van Vlissingen M, Fouchier R, de Swart R, Koopmans M, Haagmans BL. Comparative pathogenesis of COVID-19, MERS, and SARS in a nonhuman primate model. Science. 2020 May 29;368(6494):1012-1015. doi: 10.1126/science.abb7314. Epub 2020 Apr 17. PMID 32303590
- [Background] Zou L, Ruan F, Huang M, Liang L, Huang H, Hong Z, Yu J, Kang M, Song Y, Xia J, Guo Q, Song T, He J, Yen HL, Peiris M, Wu J. SARS-CoV-2 Viral Load in Upper Respiratory Specimens of Infected Patients. N Engl J Med. 2020 Mar 19;382(12):1177-1179. doi: 10.1056/NEJMc2001737. Epub 2020 Feb 19. No abstract available. PMID 32074444
- [Background] Meng X, Deng Y, Dai Z, Meng Z. COVID-19 and anosmia: A review based on up-to-date knowledge. Am J Otolaryngol. 2020 Sep-Oct;41(5):102581. doi: 10.1016/j.amjoto.2020.102581. Epub 2020 Jun 2. PMID 32563019
- [Background] Baig AM, Khaleeq A, Ali U, Syeda H. Evidence of the COVID-19 Virus Targeting the CNS: Tissue Distribution, Host-Virus Interaction, and Proposed Neurotropic Mechanisms. ACS Chem Neurosci. 2020 Apr 1;11(7):995-998. doi: 10.1021/acschemneuro.0c00122. Epub 2020 Mar 13. PMID 32167747
- [Background] Brann DH, Tsukahara T, Weinreb C, Lipovsek M, Van den Berge K, Gong B, Chance R, Macaulay IC, Chou HJ, Fletcher RB, Das D, Street K, de Bezieux HR, Choi YG, Risso D, Dudoit S, Purdom E, Mill J, Hachem RA, Matsunami H, Logan DW, Goldstein BJ, Grubb MS, Ngai J, Datta SR. Non-neuronal expression of SARS-CoV-2 entry genes in the olfactory system suggests mechanisms underlying COVID-19-associated anosmia. Sci Adv. 2020 Jul 31;6(31):eabc5801. doi: 10.1126/sciadv.abc5801. Epub 2020 Jul 24. PMID 32937591
- [Background] Morbini P, Benazzo M, Verga L, Pagella FG, Mojoli F, Bruno R, Marena C. Ultrastructural Evidence of Direct Viral Damage to the Olfactory Complex in Patients Testing Positive for SARS-CoV-2. JAMA Otolaryngol Head Neck Surg. 2020 Oct 1;146(10):972-973. doi: 10.1001/jamaoto.2020.2366. No abstract available. PMID 32790835
- [Background] Politi LS, Salsano E, Grimaldi M. Magnetic Resonance Imaging Alteration of the Brain in a Patient With Coronavirus Disease 2019 (COVID-19) and Anosmia. JAMA Neurol. 2020 Aug 1;77(8):1028-1029. doi: 10.1001/jamaneurol.2020.2125. No abstract available. PMID 32469400
- [Background] Wilson DA, Best AR, Sullivan RM. Plasticity in the olfactory system: lessons for the neurobiology of memory. Neuroscientist. 2004 Dec;10(6):513-24. doi: 10.1177/1073858404267048. PMID 15534037
- [Background] Kollndorfer K, Kowalczyk K, Hoche E, Mueller CA, Pollak M, Trattnig S, Schopf V. Recovery of olfactory function induces neuroplasticity effects in patients with smell loss. Neural Plast. 2014;2014:140419. doi: 10.1155/2014/140419. Epub 2014 Dec 3. PMID 25544900
- [Background] Giacomelli A, Pezzati L, Conti F, Bernacchia D, Siano M, Oreni L, Rusconi S, Gervasoni C, Ridolfo AL, Rizzardini G, Antinori S, Galli M. Self-reported Olfactory and Taste Disorders in Patients With Severe Acute Respiratory Coronavirus 2 Infection: A Cross-sectional Study. Clin Infect Dis. 2020 Jul 28;71(15):889-890. doi: 10.1093/cid/ciaa330. No abstract available. PMID 32215618
- [Background] Lechien JR, Barillari MR, Jouffe L, Saussez S. Anosmia Is a Key Symptom of COVID-19 Infection and Should Be Used as a Diagnostic Tool. Ear Nose Throat J. 2020 Nov;99(9):577-578. doi: 10.1177/0145561320925191. Epub 2020 May 21. PMID 32436441
- [Background] Moein ST, Hashemian SM, Mansourafshar B, Khorram-Tousi A, Tabarsi P, Doty RL. Smell dysfunction: a biomarker for COVID-19. Int Forum Allergy Rhinol. 2020 Aug;10(8):944-950. doi: 10.1002/alr.22587. Epub 2020 Jun 18. PMID 32301284
- [Background] Spinato G, Fabbris C, Polesel J, Cazzador D, Borsetto D, Hopkins C, Boscolo-Rizzo P. Alterations in Smell or Taste in Mildly Symptomatic Outpatients With SARS-CoV-2 Infection. JAMA. 2020 May 26;323(20):2089-2090. doi: 10.1001/jama.2020.6771. PMID 32320008
- [Background] Menni C, Valdes AM, Freidin MB, Sudre CH, Nguyen LH, Drew DA, Ganesh S, Varsavsky T, Cardoso MJ, El-Sayed Moustafa JS, Visconti A, Hysi P, Bowyer RCE, Mangino M, Falchi M, Wolf J, Ourselin S, Chan AT, Steves CJ, Spector TD. Real-time tracking of self-reported symptoms to predict potential COVID-19. Nat Med. 2020 Jul;26(7):1037-1040. doi: 10.1038/s41591-020-0916-2. Epub 2020 May 11. PMID 32393804
- [Background] Boscolo-Rizzo P, Borsetto D, Fabbris C, Spinato G, Frezza D, Menegaldo A, Mularoni F, Gaudioso P, Cazzador D, Marciani S, Frasconi S, Ferraro M, Berro C, Varago C, Nicolai P, Tirelli G, Da Mosto MC, Obholzer R, Rigoli R, Polesel J, Hopkins C. Evolution of Altered Sense of Smell or Taste in Patients With Mildly Symptomatic COVID-19. JAMA Otolaryngol Head Neck Surg. 2020 Aug 1;146(8):729-732. doi: 10.1001/jamaoto.2020.1379. PMID 32614442
- [Background] Hendriks AP. Olfactory dysfunction. Rhinology. 1988 Dec;26(4):229-51. PMID 3070710
- [Background] Reden J, Mueller A, Mueller C, Konstantinidis I, Frasnelli J, Landis BN, Hummel T. Recovery of olfactory function following closed head injury or infections of the upper respiratory tract. Arch Otolaryngol Head Neck Surg. 2006 Mar;132(3):265-9. doi: 10.1001/archotol.132.3.265. PMID 16549746
- [Background] Lechien JR, Chiesa-Estomba CM, Beckers E, Mustin V, Ducarme M, Journe F, Marchant A, Jouffe L, Barillari MR, Cammaroto G, Circiu MP, Hans S, Saussez S. Prevalence and 6-month recovery of olfactory dysfunction: a multicentre study of 1363 COVID-19 patients. J Intern Med. 2021 Aug;290(2):451-461. doi: 10.1111/joim.13209. Epub 2021 Jan 5. PMID 33403772
- [Background] Renaud M, Thibault C, Le Normand F, Mcdonald EG, Gallix B, Debry C, Venkatasamy A. Clinical Outcomes for Patients With Anosmia 1 Year After COVID-19 Diagnosis. JAMA Netw Open. 2021 Jun 1;4(6):e2115352. doi: 10.1001/jamanetworkopen.2021.15352. PMID 34165581
- [Background] Whitcroft KL, Hummel T. Olfactory Dysfunction in COVID-19: Diagnosis and Management. JAMA. 2020 Jun 23;323(24):2512-2514. doi: 10.1001/jama.2020.8391. No abstract available. PMID 32432682
- [Background] Rawal S, Hoffman HJ, Bainbridge KE, Huedo-Medina TB, Duffy VB. Prevalence and Risk Factors of Self-Reported Smell and Taste Alterations: Results from the 2011-2012 US National Health and Nutrition Examination Survey (NHANES). Chem Senses. 2016 Jan;41(1):69-76. doi: 10.1093/chemse/bjv057. Epub 2015 Oct 20. PMID 26487703
- [Background] Reden J, Maroldt H, Fritz A, Zahnert T, Hummel T. A study on the prognostic significance of qualitative olfactory dysfunction. Eur Arch Otorhinolaryngol. 2007 Feb;264(2):139-44. doi: 10.1007/s00405-006-0157-0. Epub 2006 Sep 28. PMID 17006637
- [Background] Graziadei PP, Levine RR, Monti Graziadei GA. Plasticity of connections of the olfactory sensory neuron: regeneration into the forebrain following bulbectomy in the neonatal mouse. Neuroscience. 1979;4(6):713-27. doi: 10.1016/0306-4522(79)90002-2. No abstract available. PMID 481748
- [Background] Seiden AM, Duncan HJ. The diagnosis of a conductive olfactory loss. Laryngoscope. 2001 Jan;111(1):9-14. doi: 10.1097/00005537-200101000-00002. PMID 11192906
- [Background] Saniasiaya J, Narayanan P. Parosmia post COVID-19: an unpleasant manifestation of long COVID syndrome. Postgrad Med J. 2021 Mar 31:postgradmedj-2021-139855. doi: 10.1136/postgradmedj-2021-139855. Online ahead of print. No abstract available. PMID 33790036
- [Background] Cavazzana A, Larsson M, Munch M, Hahner A, Hummel T. Postinfectious olfactory loss: A retrospective study on 791 patients. Laryngoscope. 2018 Jan;128(1):10-15. doi: 10.1002/lary.26606. Epub 2017 May 29. PMID 28556265
- [Background] Kim DH, Kim SW, Hwang SH, Kim BG, Kang JM, Cho JH, Park YJ, Kim SW. Prognosis of Olfactory Dysfunction according to Etiology and Timing of Treatment. Otolaryngol Head Neck Surg. 2017 Feb;156(2):371-377. doi: 10.1177/0194599816679952. Epub 2016 Dec 20. PMID 28145844
- [Background] Schriever VA, Merkonidis C, Gupta N, Hummel C, Hummel T. Treatment of smell loss with systemic methylprednisolone. Rhinology. 2012 Sep;50(3):284-9. doi: 10.4193/Rhino.11.207. PMID 22888485
- [Background] Seo BS, Lee HJ, Mo JH, Lee CH, Rhee CS, Kim JW. Treatment of postviral olfactory loss with glucocorticoids, Ginkgo biloba, and mometasone nasal spray. Arch Otolaryngol Head Neck Surg. 2009 Oct;135(10):1000-4. doi: 10.1001/archoto.2009.141. PMID 19841338
- [Background] Blomqvist EH, Lundblad L, Bergstedt H, Stjarne P. Placebo-controlled, randomized, double-blind study evaluating the efficacy of fluticasone propionate nasal spray for the treatment of patients with hyposmia/anosmia. Acta Otolaryngol. 2003 Sep;123(7):862-8. doi: 10.1080/00016480310002140. PMID 14575403
- [Background] Friedman M, Hamilton C, Samuelson CG, Maley A, Wilson MN, Venkatesan TK, Joseph NJ. Dead Sea salt irrigations vs saline irrigations with nasal steroids for symptomatic treatment of chronic rhinosinusitis: a randomized, prospective double-blind study. Int Forum Allergy Rhinol. 2012 May-Jun;2(3):252-7. doi: 10.1002/alr.21003. Epub 2012 Feb 15. PMID 22337474
- [Background] Yan CH, Overdevest JB, Patel ZM. Therapeutic use of steroids in non-chronic rhinosinusitis olfactory dysfunction: a systematic evidence-based review with recommendations. Int Forum Allergy Rhinol. 2019 Feb;9(2):165-176. doi: 10.1002/alr.22240. Epub 2018 Nov 24. PMID 30472771
- [Background] Nguyen TP, Patel ZM. Budesonide irrigation with olfactory training improves outcomes compared with olfactory training alone in patients with olfactory loss. Int Forum Allergy Rhinol. 2018 Sep;8(9):977-981. doi: 10.1002/alr.22140. Epub 2018 Jun 14. PMID 29901865
- [Background] Barnes PJ. Theophylline. Pharmaceuticals (Basel). 2010 Mar 18;3(3):725-747. doi: 10.3390/ph3030725. PMID 27713276
- [Background] Tomita K, Chikumi H, Tokuyasu H, Yajima H, Hitsuda Y, Matsumoto Y, Sasaki T. Functional assay of NF-kappaB translocation into nuclei by laser scanning cytometry: inhibitory effect by dexamethasone or theophylline. Naunyn Schmiedebergs Arch Pharmacol. 1999 Apr;359(4):249-55. doi: 10.1007/pl00005349. PMID 10344522
- [Background] Henkin RI, Schultz M, Minnick-Poppe L. Intranasal theophylline treatment of hyposmia and hypogeusia: a pilot study. Arch Otolaryngol Head Neck Surg. 2012 Nov;138(11):1064-70. doi: 10.1001/2013.jamaoto.342. PMID 23165381
- [Background] Moon C, Simpson PJ, Tu Y, Cho H, Ronnett GV. Regulation of intracellular cyclic GMP levels in olfactory sensory neurons. J Neurochem. 2005 Oct;95(1):200-9. doi: 10.1111/j.1471-4159.2005.03356.x. PMID 16181424
- [Background] Pace U, Hanski E, Salomon Y, Lancet D. Odorant-sensitive adenylate cyclase may mediate olfactory reception. Nature. 1985 Jul 18-24;316(6025):255-8. doi: 10.1038/316255a0. PMID 3927168
- [Background] Ronnett GV, Parfitt DJ, Hester LD, Snyder SH. Odorant-sensitive adenylate cyclase: rapid, potent activation and desensitization in primary olfactory neuronal cultures. Proc Natl Acad Sci U S A. 1991 Mar 15;88(6):2366-9. doi: 10.1073/pnas.88.6.2366. PMID 2006174
- [Background] Anholt RR. Molecular neurobiology of olfaction. Crit Rev Neurobiol. 1993;7(1):1-22. PMID 8467526
- [Background] Neumann S, Bradke F, Tessier-Lavigne M, Basbaum AI. Regeneration of sensory axons within the injured spinal cord induced by intraganglionic cAMP elevation. Neuron. 2002 Jun 13;34(6):885-93. doi: 10.1016/s0896-6273(02)00702-x. PMID 12086637
- [Background] Henkin RI, Velicu I. cAMP and cGMP in nasal mucus: relationships to taste and smell dysfunction, gender and age. Clin Invest Med. 2008;31(2):E71-7. doi: 10.25011/cim.v31i2.3366. PMID 18377763
- [Background] Henkin RI, Velicu I. cAMP and cGMP in nasal mucus related to severity of smell loss in patients with smell dysfunction. Clin Invest Med. 2008;31(2):E78-84. doi: 10.25011/cim.v31i2.3367. PMID 18377764
- [Background] Henkin RI, Velicu I, Schmidt L. An open-label controlled trial of theophylline for treatment of patients with hyposmia. Am J Med Sci. 2009 Jun;337(6):396-406. doi: 10.1097/MAJ.0b013e3181914a97. PMID 19359985
- [Background] Levy LM, Henkin RI, Lin CS, Hutter A, Schellinger D. Increased brain activation in response to odors in patients with hyposmia after theophylline treatment demonstrated by fMRI. J Comput Assist Tomogr. 1998 Sep-Oct;22(5):760-70. doi: 10.1097/00004728-199809000-00019. PMID 9754114
- [Background] Balmer JE, Blomhoff R. Gene expression regulation by retinoic acid. J Lipid Res. 2002 Nov;43(11):1773-808. doi: 10.1194/jlr.r100015-jlr200. PMID 12401878
- [Background] Rawson NE, LaMantia AS. A speculative essay on retinoic acid regulation of neural stem cells in the developing and aging olfactory system. Exp Gerontol. 2007 Jan-Feb;42(1-2):46-53. doi: 10.1016/j.exger.2006.05.021. Epub 2006 Jul 24. PMID 16860961
- [Background] Hummel T, Whitcroft KL, Rueter G, Haehner A. Intranasal vitamin A is beneficial in post-infectious olfactory loss. Eur Arch Otorhinolaryngol. 2017 Jul;274(7):2819-2825. doi: 10.1007/s00405-017-4576-x. Epub 2017 Apr 22. PMID 28434127
- [Background] Carrie I, Abellan Van Kan G, Rolland Y, Gillette-Guyonnet S, Vellas B. PUFA for prevention and treatment of dementia? Curr Pharm Des. 2009;15(36):4173-85. doi: 10.2174/138161209789909764. PMID 20041819
- [Background] Calder PC. Omega-3 fatty acids and inflammatory processes: from molecules to man. Biochem Soc Trans. 2017 Oct 15;45(5):1105-1115. doi: 10.1042/BST20160474. Epub 2017 Sep 12. PMID 28900017
- [Background] Gopinath B, Sue CM, Flood VM, Burlutsky G, Mitchell P. Dietary intakes of fats, fish and nuts and olfactory impairment in older adults. Br J Nutr. 2015 Jul;114(2):240-7. doi: 10.1017/S0007114515001257. Epub 2015 Jun 16. PMID 26079067
- [Background] Yan CH, Rathor A, Krook K, Ma Y, Rotella MR, Dodd RL, Hwang PH, Nayak JV, Oyesiku NM, DelGaudio JM, Levy JM, Wise J, Wise SK, Patel ZM. Effect of Omega-3 Supplementation in Patients With Smell Dysfunction Following Endoscopic Sellar and Parasellar Tumor Resection: A Multicenter Prospective Randomized Controlled Trial. Neurosurgery. 2020 Aug 1;87(2):E91-E98. doi: 10.1093/neuros/nyz559. PMID 31950156
- [Background] Rondanelli M, Opizzi A, Faliva M, Mozzoni M, Antoniello N, Cazzola R, Savare R, Cerutti R, Grossi E, Cestaro B. Effects of a diet integration with an oily emulsion of DHA-phospholipids containing melatonin and tryptophan in elderly patients suffering from mild cognitive impairment. Nutr Neurosci. 2012 Mar;15(2):46-54. doi: 10.1179/1476830511Y.0000000032. Epub 2011 Dec 20. PMID 22334085
- [Background] Jiang X, Finucane HK, Schumacher FR, Schmit SL, Tyrer JP, Han Y, Michailidou K, Lesseur C, Kuchenbaecker KB, Dennis J, Conti DV, Casey G, Gaudet MM, Huyghe JR, Albanes D, Aldrich MC, Andrew AS, Andrulis IL, Anton-Culver H, Antoniou AC, Antonenkova NN, Arnold SM, Aronson KJ, Arun BK, Bandera EV, Barkardottir RB, Barnes DR, Batra J, Beckmann MW, Benitez J, Benlloch S, Berchuck A, Berndt SI, Bickeboller H, Bien SA, Blomqvist C, Boccia S, Bogdanova NV, Bojesen SE, Bolla MK, Brauch H, Brenner H, Brenton JD, Brook MN, Brunet J, Brunnstrom H, Buchanan DD, Burwinkel B, Butzow R, Cadoni G, Caldes T, Caligo MA, Campbell I, Campbell PT, Cancel-Tassin G, Cannon-Albright L, Campa D, Caporaso N, Carvalho AL, Chan AT, Chang-Claude J, Chanock SJ, Chen C, Christiani DC, Claes KBM, Claessens F, Clements J, Collee JM, Correa MC, Couch FJ, Cox A, Cunningham JM, Cybulski C, Czene K, Daly MB, deFazio A, Devilee P, Diez O, Gago-Dominguez M, Donovan JL, Dork T, Duell EJ, Dunning AM, Dwek M, Eccles DM, Edlund CK, Edwards DRV, Ellberg C, Evans DG, Fasching PA, Ferris RL, Liloglou T, Figueiredo JC, Fletcher O, Fortner RT, Fostira F, Franceschi S, Friedman E, Gallinger SJ, Ganz PA, Garber J, Garcia-Saenz JA, Gayther SA, Giles GG, Godwin AK, Goldberg MS, Goldgar DE, Goode EL, Goodman MT, Goodman G, Grankvist K, Greene MH, Gronberg H, Gronwald J, Guenel P, Hakansson N, Hall P, Hamann U, Hamdy FC, Hamilton RJ, Hampe J, Haugen A, Heitz F, Herrero R, Hillemanns P, Hoffmeister M, Hogdall E, Hong YC, Hopper JL, Houlston R, Hulick PJ, Hunter DJ, Huntsman DG, Idos G, Imyanitov EN, Ingles SA, Isaacs C, Jakubowska A, James P, Jenkins MA, Johansson M, Johansson M, John EM, Joshi AD, Kaneva R, Karlan BY, Kelemen LE, Kuhl T, Khaw KT, Khusnutdinova E, Kibel AS, Kiemeney LA, Kim J, Kjaer SK, Knight JA, Kogevinas M, Kote-Jarai Z, Koutros S, Kristensen VN, Kupryjanczyk J, Lacko M, Lam S, Lambrechts D, Landi MT, Lazarus P, Le ND, Lee E, Lejbkowicz F, Lenz HJ, Leslie G, Lessel D, Lester J, Levine DA, Li L, Li CI, Lindblom A, Lindor NM, Liu G, Loupakis F, Lubinski J, Maehle L, Maier C, Mannermaa A, Marchand LL, Margolin S, May T, McGuffog L, Meindl A, Middha P, Miller A, Milne RL, MacInnis RJ, Modugno F, Montagna M, Moreno V, Moysich KB, Mucci L, Muir K, Mulligan AM, Nathanson KL, Neal DE, Ness AR, Neuhausen SL, Nevanlinna H, Newcomb PA, Newcomb LF, Nielsen FC, Nikitina-Zake L, Nordestgaard BG, Nussbaum RL, Offit K, Olah E, Olama AAA, Olopade OI, Olshan AF, Olsson H, Osorio A, Pandha H, Park JY, Pashayan N, Parsons MT, Pejovic T, Penney KL, Peters WHM, Phelan CM, Phipps AI, Plaseska-Karanfilska D, Pring M, Prokofyeva D, Radice P, Stefansson K, Ramus SJ, Raskin L, Rennert G, Rennert HS, van Rensburg EJ, Riggan MJ, Risch HA, Risch A, Roobol MJ, Rosenstein BS, Rossing MA, De Ruyck K, Saloustros E, Sandler DP, Sawyer EJ, Schabath MB, Schleutker J, Schmidt MK, Setiawan VW, Shen H, Siegel EM, Sieh W, Singer CF, Slattery ML, Sorensen KD, Southey MC, Spurdle AB, Stanford JL, Stevens VL, Stintzing S, Stone J, Sundfeldt K, Sutphen R, Swerdlow AJ, Tajara EH, Tangen CM, Tardon A, Taylor JA, Teare MD, Teixeira MR, Terry MB, Terry KL, Thibodeau SN, Thomassen M, Bjorge L, Tischkowitz M, Toland AE, Torres D, Townsend PA, Travis RC, Tung N, Tworoger SS, Ulrich CM, Usmani N, Vachon CM, Van Nieuwenhuysen E, Vega A, Aguado-Barrera ME, Wang Q, Webb PM, Weinberg CR, Weinstein S, Weissler MC, Weitzel JN, West CML, White E, Whittemore AS, Wichmann HE, Wiklund F, Winqvist R, Wolk A, Woll P, Woods M, Wu AH, Wu X, Yannoukakos D, Zheng W, Zienolddiny S, Ziogas A, Zorn KK, Lane JM, Saxena R, Thomas D, Hung RJ, Diergaarde B, McKay J, Peters U, Hsu L, Garcia-Closas M, Eeles RA, Chenevix-Trench G, Brennan PJ, Haiman CA, Simard J, Easton DF, Gruber SB, Pharoah PDP, Price AL, Pasaniuc B, Amos CI, Kraft P, Lindstrom S. Shared heritability and functional enrichment across six solid cancers. Nat Commun. 2019 Jan 25;10(1):431. doi: 10.1038/s41467-018-08054-4. PMID 30683880
- [Background] Bourrie B, Bribes E, Derocq JM, Vidal H, Casellas P. Sigma receptor ligands: applications in inflammation and oncology. Curr Opin Investig Drugs. 2004 Nov;5(11):1158-63. PMID 15573866
- [Background] Lewis R, Li J, McCormick PJ, L-H Huang C, Jeevaratnam K. Is the sigma-1 receptor a potential pharmacological target for cardiac pathologies? A systematic review. Int J Cardiol Heart Vasc. 2019 Dec 28;26:100449. doi: 10.1016/j.ijcha.2019.100449. eCollection 2020 Feb. PMID 31909177
- [Background] Oxombre B, Lee-Chang C, Duhamel A, Toussaint M, Giroux M, Donnier-Marechal M, Carato P, Lefranc D, Zephir H, Prin L, Melnyk P, Vermersch P. High-affinity sigma1 protein agonist reduces clinical and pathological signs of experimental autoimmune encephalomyelitis. Br J Pharmacol. 2015 Apr;172(7):1769-82. doi: 10.1111/bph.13037. Epub 2015 Feb 10. PMID 25521311
- [Background] Nishimura T, Ishima T, Iyo M, Hashimoto K. Potentiation of nerve growth factor-induced neurite outgrowth by fluvoxamine: role of sigma-1 receptors, IP3 receptors and cellular signaling pathways. PLoS One. 2008 Jul 2;3(7):e2558. doi: 10.1371/journal.pone.0002558. PMID 18596927
- [Background] Hashimoto K. Sigma-1 receptor chaperone and brain-derived neurotrophic factor: emerging links between cardiovascular disease and depression. Prog Neurobiol. 2013 Jan;100:15-29. doi: 10.1016/j.pneurobio.2012.09.001. Epub 2012 Oct 5. PMID 23044468
- [Background] Ishima T, Fujita Y, Hashimoto K. Interaction of new antidepressants with sigma-1 receptor chaperones and their potentiation of neurite outgrowth in PC12 cells. Eur J Pharmacol. 2014 Mar 15;727:167-73. doi: 10.1016/j.ejphar.2014.01.064. Epub 2014 Feb 5. PMID 24508523
- [Background] Hashimoto K. Activation of sigma-1 receptor chaperone in the treatment of neuropsychiatric diseases and its clinical implication. J Pharmacol Sci. 2015 Jan;127(1):6-9. doi: 10.1016/j.jphs.2014.11.010. Epub 2014 Dec 4. PMID 25704012
- [Background] Cobos EJ, Entrena JM, Nieto FR, Cendan CM, Del Pozo E. Pharmacology and therapeutic potential of sigma(1) receptor ligands. Curr Neuropharmacol. 2008 Dec;6(4):344-66. doi: 10.2174/157015908787386113. PMID 19587856
- [Background] Hallifax D, Houston JB. Saturable uptake of lipophilic amine drugs into isolated hepatocytes: mechanisms and consequences for quantitative clearance prediction. Drug Metab Dispos. 2007 Aug;35(8):1325-32. doi: 10.1124/dmd.107.015131. Epub 2007 Apr 30. PMID 17470525
- [Background] Sukhatme VP, Reiersen AM, Vayttaden SJ, Sukhatme VV. Fluvoxamine: A Review of Its Mechanism of Action and Its Role in COVID-19. Front Pharmacol. 2021 Apr 20;12:652688. doi: 10.3389/fphar.2021.652688. eCollection 2021. PMID 33959018
- [Background] Lenze EJ, Mattar C, Zorumski CF, Stevens A, Schweiger J, Nicol GE, Miller JP, Yang L, Yingling M, Avidan MS, Reiersen AM. Fluvoxamine vs Placebo and Clinical Deterioration in Outpatients With Symptomatic COVID-19: A Randomized Clinical Trial. JAMA. 2020 Dec 8;324(22):2292-2300. doi: 10.1001/jama.2020.22760. PMID 33180097
- [Background] Reis G, Dos Santos Moreira-Silva EA, Silva DCM, Thabane L, Milagres AC, Ferreira TS, Dos Santos CVQ, de Souza Campos VH, Nogueira AMR, de Almeida APFG, Callegari ED, de Figueiredo Neto AD, Savassi LCM, Simplicio MIC, Ribeiro LB, Oliveira R, Harari O, Forrest JI, Ruton H, Sprague S, McKay P, Glushchenko AV, Rayner CR, Lenze EJ, Reiersen AM, Guyatt GH, Mills EJ; TOGETHER investigators. Effect of early treatment with fluvoxamine on risk of emergency care and hospitalisation among patients with COVID-19: the TOGETHER randomised, platform clinical trial. Lancet Glob Health. 2022 Jan;10(1):e42-e51. doi: 10.1016/S2214-109X(21)00448-4. Epub 2021 Oct 28. PMID 34717820
- [Background] Kroenke K, Spitzer RL, Williams JB. The PHQ-9: validity of a brief depression severity measure. J Gen Intern Med. 2001 Sep;16(9):606-13. doi: 10.1046/j.1525-1497.2001.016009606.x. PMID 11556941
- [Background] Dunlop BW, Gray J, Rapaport MH. Transdiagnostic Clinical Global Impression Scoring for Routine Clinical Settings. Behav Sci (Basel). 2017 Jun 27;7(3):40. doi: 10.3390/bs7030040. PMID 28653978
- [Background] Doty RL, Shaman P, Kimmelman CP, Dann MS. University of Pennsylvania Smell Identification Test: a rapid quantitative olfactory function test for the clinic. Laryngoscope. 1984 Feb;94(2 Pt 1):176-8. doi: 10.1288/00005537-198402000-00004. PMID 6694486
- [Background] Ware JE Jr, Sherbourne CD. The MOS 36-item short-form health survey (SF-36). I. Conceptual framework and item selection. Med Care. 1992 Jun;30(6):473-83. PMID 1593914
- [Background] Henry JA. Overdose and safety with fluvoxamine. Int Clin Psychopharmacol. 1991 Dec;6 Suppl 3:41-5; discussion 45-7. doi: 10.1097/00004850-199112003-00004. PMID 1806634
- [Background] Kharasch ED, Neiner A, Kraus K, Blood J, Stevens A, Schweiger J, Miller JP, Lenze EJ. Bioequivalence and Therapeutic Equivalence of Generic and Brand Bupropion in Adults With Major Depression: A Randomized Clinical Trial. Clin Pharmacol Ther. 2019 May;105(5):1164-1174. doi: 10.1002/cpt.1309. Epub 2019 Jan 18. PMID 30460996
- [Background] Lenze EJ, Stevens A, Waring JD, Pham VT, Haddad R, Shimony J, Miller JP, Bowie CR. Augmenting Computerized Cognitive Training With Vortioxetine for Age-Related Cognitive Decline: A Randomized Controlled Trial. Am J Psychiatry. 2020 Jun 1;177(6):548-555. doi: 10.1176/appi.ajp.2019.19050561. Epub 2020 Mar 26. PMID 32212856
- [Background] Christensen M, Tybring G, Mihara K, Yasui-Furokori N, Carrillo JA, Ramos SI, Andersson K, Dahl ML, Bertilsson L. Low daily 10-mg and 20-mg doses of fluvoxamine inhibit the metabolism of both caffeine (cytochrome P4501A2) and omeprazole (cytochrome P4502C19). Clin Pharmacol Ther. 2002 Mar;71(3):141-52. doi: 10.1067/mcp.2002.121788. PMID 11907488
- [Background] Budha NR, Ji T, Musib L, Eppler S, Dresser M, Chen Y, Jin JY. Evaluation of Cytochrome P450 3A4-Mediated Drug-Drug Interaction Potential for Cobimetinib Using Physiologically Based Pharmacokinetic Modeling and Simulation. Clin Pharmacokinet. 2016 Nov;55(11):1435-1445. doi: 10.1007/s40262-016-0412-5. PMID 27225997
- [Background] Vezmar S, Miljkovic B, Vucicevic K, Timotijevic I, Prostran M, Todorovic Z, Pokrajac M. Pharmacokinetics and efficacy of fluvoxamine and amitriptyline in depression. J Pharmacol Sci. 2009 May;110(1):98-104. doi: 10.1254/jphs.09013fp. PMID 19444001
- [Background] Gebara MA, Shea ML, Lipsey KL, Teitelbaum SL, Civitelli R, Muller DJ, Reynolds CF 3rd, Mulsant BH, Lenze EJ. Depression, antidepressants, and bone health in older adults: a systematic review. J Am Geriatr Soc. 2014 Aug;62(8):1434-41. doi: 10.1111/jgs.12945. Epub 2014 Jul 15. PMID 25039259
- [Background] Dixon AE, Kaminsky DA, Holbrook JT, Wise RA, Shade DM, Irvin CG. Allergic rhinitis and sinusitis in asthma: differential effects on symptoms and pulmonary function. Chest. 2006 Aug;130(2):429-35. doi: 10.1378/chest.130.2.429. PMID 16899841
- [Background] Gebara MA, Lipsey KL, Karp JF, Nash MC, Iaboni A, Lenze EJ. Cause or Effect? Selective Serotonin Reuptake Inhibitors and Falls in Older Adults: A Systematic Review. Am J Geriatr Psychiatry. 2015 Oct;23(10):1016-28. doi: 10.1016/j.jagp.2014.11.004. Epub 2014 Nov 25. PMID 25586602
- See also: article discussing early symptoms of Covid-19 infection — http://www.medrxiv.org/content/10.1101/2020.04.05.20048421v1
- See also: American Academy of Otolaryngology - Head and Neck Surgery — http://www.entnet.org/content/aao-hns-anosmia-hyposmia-and-dysgeusia-symptoms-coronavirus-disease
- See also: ENT UK site discussing loss of smell as a covid-19 early symptom — http://www.google.com/url?sa=t&rct=j&q=&esrc=s&source=web&cd=1&ved=2ahUKEwiIy9bQ6cToAhURMawKHW5LB9UQFjAAegQIBBAB&url=https%3A%2F%2Fwww.entuk.org%2Floss-sense-smell-marker-covid-19-infection&usg=AOvVaw0W88Tj7ToIsMSc1DChCUEy
- See also: article discussing the Depression Anxiety & Stress Scale published by University of Wisconsin - Madison — http://arc.psych.wisc.edu/self-report/depression-anxiety-stress-scale-21-dass21/
- See also: article discussing the ECDEU Assessment Manual published in national catalogue — http://catalogue.nla.gov.au/Record/1010635
- Available data/document: Clinical Study Report: 10.7599/hmr.2014.34.3.107 — http://www.researchgate.net/publication/271283284_Clinical_Diagnosis_and_Treatment_of_Olfactory_Dysfunction — Research article published in Hanyang Medical Reviews discussing diagnosis and treatment of olfactory dysfunction